CLINICAL TRIAL: NCT05989373
Title: Scratch Collapse Test: Prospective, Objective, Multi Multicenter
Brief Title: Objective Evaluation of the Scratch Collapse Test With Dynamometer, a Prospective Multicenter Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Principal Investigator, Benjamin DEGEORGE, Principal investigator, Clinique Saint Jean, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01972-41
Record Dates: First submitted 2023-05-31; First posted 2023-08-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Carpal Tunnel Syndrome; Ulnar Nerve Compression
MeSH Terms: conditions — Carpal Tunnel Syndrome; Ulnar Nerve Compression Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nerve stimulation (Experimental): The test in currently used to search for a nerv compression
  Interventions: Diagnostic Test: Scratch collapse test

INTERVENTIONS:
Diagnostic Test: Scratch collapse test — Scratch test performed by the surgeon but with a dynamometer

SUMMARY:
Carpal tunnel syndrome and compression of the ulnar nerve at the elbow are common pathologies, which are treated surgically.

Diagnosis is usually based on an electromyogram (EMG), as well as symptomatology, etiology of typical symptoms and an evocative clinical examination. Provocative tests performed in consultation include the Tinel and Phalen sign for the carpal tunnel, and the Tinel and prolonged flexion sign for the ulnar nerve at the elbow.

The Scratch Collapse Test (SCT) has recently emerged as a new provocation test to help diagnose nerve compression in the upper limb.

This non-invasive, pain-free test looks for a reduction in the force of external rotation of the shoulder by applying resistance (the doctor's arm), before and then after a sensory stimulus by "scratching" the area of compression. Nevertheless, this test remains controversial and not based on objective measurements.

Our aim is therefore to assess shoulder external rotation force, and thus TBS, objectively with a dynamometer, before and after stimulation in cases of median nerve compression syndrome at the carpal tunnel and ulnar nerve compression syndrome at the elbow, when these are clinically and electromyographically proven.

This test has already been studied in the literature, but the results in terms of sensitivity and specificity are highly disparate. One study has already published negative results on the subject, with the limitation that the trial was monocentric.

Through this multicenter study, principal investigator wish to highlight the very probable subjectivity of the SCT when it is performed. As the resistance is applied by the physician's arm, the investigator cannot determine the force applied against the patient, unlike with a measurement object. The principal investigator expects this study to refute the notion that external shoulder rotation force decreases after trigger zone stimulation in cases of proven nerve compression syndrome.

The results of this study will thus make it possible to discontinue the use of this technique if it does not help in the diagnosis of compression.

The literature shows a lack of prospective, objective studies involving a large number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated or entitled to a social security plan
* Patient who has received informed information about the study
* Patient of legal age
* Patient with ulnar nerve or carpal tunnel compression confirmed by EMG during preoperative consultation

Exclusion Criteria:

* Recurrence of nerve compression
* Any history that may affect arm sensitivity
* Infra-electromyographic nerve compression syndrome (pure ulnar nerve instability)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Variation in the force of external rotation of the elbow | Inclusion day
  measurement taken before the test and the measurement taken immediately after nerve stimulation according to the SCT. The force is measured with a dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique St Jean sud de france, Saint-Jean-de-Védas, France

IPD SHARING:
Plan to Share IPD: No